CLINICAL TRIAL: NCT03053921
Title: Treatment of Gingival Recession Using a Coronally Advanced Flap Procedure With or Without Placental Membrane
Brief Title: Placental Membrane for Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Meenakshi Ammal Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MADC/IRB/2015/94
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-01

CONDITIONS: Gingival Recession
Keywords: gingival recession; Zuchellis technique,; placental membrane
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recession coverage (Placebo Comparator): 30 recession defects treated with Zucchelli's technique.
  Interventions: Procedure: recession coverage
- recession coverage and membrane (Active Comparator): 30 recession defects treated with Zucchelli's technique along with placental membrane.
  Interventions: Procedure: recession coverage and membrane

INTERVENTIONS:
Procedure: recession coverage — recession coverage done using Zuchellis technique
  Other Names: root coverage technique
  Arms: recession coverage
Procedure: recession coverage and membrane — recession coverage done using Zuchellis technique with placental membrane
  Other Names: root coverage technique with membrane
  Arms: recession coverage and membrane

SUMMARY:
Aim of the study was to evaluate the clinical efficacy of placental membrane with coronally advanced flap in covering single and multiple Miller's class I and II gingival recession defects.

DETAILED DESCRIPTION:
STUDY DESIGN A total number of 60 teeth in 15 subjects were selected. Patients with bilateral Miller's class I and II gingival recession defects in the maxillary or mandibular anterior and premolar region were selected and divided into two groups using a split mouth design.

GroupI (Control) -30 recession defects treated with coronally advanced flap alone, using Zucchelli's technique.

Group II (Test) - 30 recession defects treated with coronally advanced flap, using Zucchelli's technique along with placental membrane.

.

CLINICAL PARAMETERS:

1. Probing Pocket Depth(PPD)
2. Clinical Attachment Level(CAL)
3. Height of Gingival Recession(HGR)
4. Width of Gingival Recession(WGR)
5. Width of Keratinized Gingiva(WKG) The clinical parameters were assessed & recorded on 0 day, 90th day and 180th day

ELIGIBILITY:
Inclusion Criteria:

1. Patients within the age group 23 to 55 years
2. Bilateral, upper or lower, Miller's class I and Class II gingival recession defects confined to the anterior and premolar region.
3. Presence of identifiable cemento-enamel junction
4. Presence of keratinized tissue apical to the exposed root

Exclusion Criteria:

1. Systemic complications
2. Occlusal interferences
3. Any contraindication for periodontal surgery and taking medication which are known to interfere with periodontal tissue health or healing
4. Previous periodontal surgery on the involved site
5. Smokers
6. Pregnant and lactating mothers

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Height of Gingival recession | 6 months
  The height of gingival recession was measured from the cemento-enamel junction to the gingival margin using Williams periodontal probe

SECONDARY OUTCOMES:
Clinical attachment level | Baseline and 6 months
  Clinical attachment level is measured as the distance between a fixed point on the crown such as cementoenamel junction to the base of the pocket using williams periodontal probe
Width of Keratinized Gingiva | Baseline and 6 months
  It is measured as the distance from the gingival margin to the mucogingival junction using williams periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Sarah George, BDS, Principal Investigator — Meenakshi Ammal Dental College and Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Mele M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Coronally advanced flap with and without vertical releasing incisions for the treatment of multiple gingival recessions: a comparative controlled randomized clinical trial. J Periodontol. 2009 Jul;80(7):1083-94. doi: 10.1902/jop.2009.090041. PMID 19563288
- [Background] Chakraborthy S, Sambashivaiah S, Kulal R, Bilchodmath S. Amnion and Chorion Allografts in Combination with Coronally Advanced Flap in the Treatment of Gingival Recession: A Clinical Study. J Clin Diagn Res. 2015 Sep;9(9):ZC98-ZC101. doi: 10.7860/JCDR/2015/12971.6572. Epub 2015 Sep 1. PMID 26501023